CLINICAL TRIAL: NCT04725968
Title: Morbimortality in Major Urgent General Surgery in the Geriatric Patient. Observational Study of Retrospective Cohort.
Brief Title: Morbimortality in Major Urgent General Surgery in the Geriatric Patient.
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CGM-2020-108
Record Dates: First submitted 2021-01-16; First posted 2021-01-27 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Surgery--Complications; Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Urgent major general surgery — All geriatric patients (75 years and over) going under urgent major general surgery during 2018 in our centre

SUMMARY:
Retrospective observational cohort study of geriatric patients operated of urgent major general surgery in our centre during 2018.

Our principal goals are:

1. To evaluate the incidence of post operation complications and its severity (defined by the Claiven-Dindo scale)
2. To evaluate the mortality: global mortality and mortality after: 30 days, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Surgeries on the small and / or large bowel with or without intestinal resection, total colectomies, exploratory laparotomies

Exclusion Criteria:

* Polytraumatic patient, reoperations (for any cause) of scheduled and urgent surgeries

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All the geriatric patients operated of urgent major general surgery in our centre during 2018.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of complications | 30 days after surgery
  Evaluate the incidence of post operation complications and its severity (defined by the Claiven-Dindo scale).
Mortality rate | 1 year
  Global mortality and mortality after: 30 days, 6 months and 1 year.

SECONDARY OUTCOMES:
Days of admission | 30 days after surgery
days in ICU/Reanimation | 30 days after surgery
NELA Risk Score | pre-surgery
  "National Emergency Laparotomy Audit" % of death
NSQUIP Risk Score | pre-surgery
  "American College of Surgeons National Surgical Quality Improvement Program": % of death

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain